CLINICAL TRIAL: NCT01613404
Title: A Prospective, Observational, Randomized Comparative Study of Case Managed Versus Non-case Managed Initiation of Hemodialysis
Brief Title: An Observational Study of Case Managed Versus Non-case Managed Initiation of Hemodialysis
Acronym: PROSTARRT
Status: Completed | Type: Observational
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016009; EPO-ANE-4080 (Other: Janssen Inc.)
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Hemodialysis; Eprex; Aranesp; ESA; Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with nurse case manager: Patients will receive a dedicated nurse case manager (intervention group) in this group.
  Interventions: Other: No intervention
- Patients with no nurse case manager: Patients will not receive nurse case manager (control group) in this group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients will be treated with approved erythropoiesis stimulating agent (Eprex or Aranesp) will be administered according to actual clinical practice according to guidance in the current approved product monographs. All patients will receive treatments that are prescribed by their physician according to actual clinical practice.

SUMMARY:
The purpose of the study is to compare the 90 day and 12 month composite end point of death (all-cause mortality) and hospitalization in incident hemodialysis patients randomized to receive support from a dedicated case manager (intervention group) versus those not receiving support from a dedicated case manager (control group).

DETAILED DESCRIPTION:
This is multicenter, prospective, observational, and randomized (the study drug is assigned by chance), 1-year study, in academic and community-based nephrology clinical practices that will examine the impact of a facility nurse case manager. In this study a group of patients guideline- based, algorithm- driven approach to hemodialysis initiation with targets (as per Canadian Society of Nephrology and/or International guidelines) will be used with facility nurse case manager and in control group same approach will be used without facility nurse case manager. Patients will be treated with any approved erythropoiesis stimulating agent for the correction of anemia, according to guidance in the current approved product monographs. All treatments will be prescribed by the physician according to actual clinical practice or standard of care for chronic kidney disease. The entire study duration for each participant will be approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who initiated hemodialysis and expected to be on hemodialysis for at least 1 year
* Patients initiating hemodialysis requiring treatment (erythropoiesis stimulating agent or red blood cell transfusion) to correct the anemia of chronic kidney disease who are receiving erythropoiesis stimulating agent treatment at study entry or patients who do not require erythropoiesis stimulating agent therapy (Hb within or above target range)
* Life expectancy should be more than 12 months

Exclusion Criteria:

* Patients contraindicated to receive erythropoiesis stimulating agent therapy (including but not limited to patients who develop pure red cell aplasia following treatment with any erythropoiesis stimulating agent )
* Patients entering the study on any other agent to increase red blood cell mass (such as androgen therapy, or investigational agents, or other non-approved erythropoiesis stimulating agent)
* Patients unwilling or unable to receive erythropoiesis stimulating agent therapy to correct the anemia of chronic kidney disease
* Patients with uncontrolled hypertension
* Patients who for any reason cannot receive adequate antithrombotic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the 90 day and 12 month composite end point of death (all-cause mortality) and hospitalization in incident hemodialysis patients of intervention group and control group | Up to 12 months
  Comparison of the 90 day and 12 month composite end point of death (all-cause mortality) and hospitalization in incident hemodialysis patients randomized to receive support from a dedicated case manager (intervention group) versus those not receiving support from a dedicated case manager (control group).

SECONDARY OUTCOMES:
Number of patients in intervention group achieving 80% of dry weight with normal blood pressure and no signs of volume overload as compared to control group | Up to 12 months
  The number of patients achieving 80% of dry weight (the amount of body mass [weight] without extra fluid [water])with normal blood pressure and no signs of volume overload in intervention group versus the control group.
Number of patients in intervention group achieving intra-dialytic weight gain (IDWG) <3Kg (based on the average over last week) as compared to control group | Up to 12 months
  The number of patients achieving 80% of intra-dialytic weight gain (IDWG) <3Kg (based on the average over last week) in intervention group versus the control group.
Number of patients in intervention group achieving hemoglobin (Hb) targeted according to guidance in the current and approved product monograph (value based on the most recent Hb result) as compared to control group | Up to 12 months
  The number of patients achieving 80% of hemoglobin (Hb) targeted according to guidance in the current and approved product monograph (value based on the most recent Hb result) in intervention group versus the control group.
Number of patients in intervention group achieving urea reduction ratio (URR) >70% (based on most recent value) as compared to control group | Up to 12 months
  The number of patients achieving 80% of urea reduction ratio (URR) >70% (based on most recent value) in intervention group versus the control group.
Number of patients achieving functioning arterio-venous fistula/arterio-venous graft (AVF/AVG) | Up to 12 months
  The number of patients achieving 80% of functioning arterio-venous fistula/arterio-venous graft (AVF/AVG) in intervention group (case managed) versus the control group (non-case managed).
Number of patients in intervention group achieving albumin >lower limit of normal (LLN) as compared to control group | Up to 12 months
  The number of patients achieving 80% of albumin >LLN (based on that center's serum albumin assay) in intervention group versus the control group.
Number of patients in intervention group achieving normal phosphate (PO4) as compared to control group | Up to 12 months
  The number of patients achieving 80% of normal phosphate (PO4) in intervention group versus the control group.
Comparison of Quality of Life scores in the intervention group and control group | Up to 12 months
  Evaluation of Quality of Life scores at baseline, 3, 6, 9 and 12 months as determined by the kidney disease quality of life (questionnaire) in the intervention group versus the control group.
Comparison of dialysis knowledge test scores in the intervention group and control group | Up to 12 months
  Dialysis Knowledge test scores at baseline, 3, 6 and 12 months in the intervention group versus the control group.
Comparison of resource utilization in the intervention group and control group | Up to 12 months
  Resource utilization will be evaluated on the basis of number and duration of medical care encounters, including surgeries, and other procedures, duration of hospitalization, medications received in hospital which are not protocol driven, outpatient medical encounters and treatments, cost of red blood cells transfusions, cost of hospitalization, and cost of renal replacement therapy.
Comparison of erythropoiesis stimulating agent (ESA) utilization patterns in the intervention group and control group | Up to 12 months
  ESA utilization patterns of such as dose adjustments, frequency of administration, length of titration phase, overall dose, and patterns of Hb control and variability, the increase of Hb from baseline, the maintenance of Hb concentration, the proportion of patients who exceed the Hb ceiling, the maximum Hb value, the rate of rise of Hb, the maximum rate of rise of Hb, and overall safety when Hb is targeted to the standard of care utilized at the participating centre in the intervention group versus the control group.
Comparison of time to AVF/AVG referral in the intervention group and control group | Up to 12 months
  Evaluation of time to AVF/AVG referral in the intervention group versus the control group.
Comparison of time to AVF/AVG surgery in the intervention group and control group | Up to 12 months
  Evaluation of time to AVF/AVG surgery referral in the intervention group versus the control group.
Comparison of time to AVF or AVG utilization in the intervention group and control group | Up to 12 months
  Evaluation of time to AVF or AVG utilization in the intervention group versus the control group.
Comparison of time to removal of central venous catheter (CVC) in the intervention group and control group | Up to 12 months
  Evaluation of time to removal of central venous catheter (CVC) in the intervention group versus the control group.
Number of participants with adverse events as measure of safety | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (14):
- Canada (14):
  - Halifax, Nova Scotia
  - Sydney, Nova Scotia
  - Kingston, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Point Claire, Quebec
  - Regina, Saskatchewan
  - Greenfield Park
  - Montreal
  - Saskatoon
  - St. John's
  - Toronto
  - Verdun